CLINICAL TRIAL: NCT01248806
Title: Validation of Low-dose Spiral CT for Early Diagnosis of Lung Cancer in a High Risk Population
Brief Title: Continuous Observation of Smoking Subject
Acronym: COSMOS
Status: Completed | Type: Observational
Sponsor: European Institute of Oncology (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Sponsor
Other Study IDs: IEO S39/100
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Subjects at High Risk of Lung Cancer Due to Smoking
Keywords: Lung nodule; Screening; Spiral low - dose computed tomography; Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Smokers or former smokers, Aged ≥ 50: Men and women current daily smokers or former smokers, Aged ≥ 50
  Interventions: Radiation: Low dose CT scan

INTERVENTIONS:
Radiation: Low dose CT scan — A low dose CT scan of the lungs is performed after the inclusion of the patient in the study and if negative for active disease, a CT scan if performed once per year for whole period of follow-up
  Other Names: High resoluzione CT scan

SUMMARY:
The purpose of this study is to offer annual low-dose spiral CT radiological examination for 5 years to 5000 volunteers from the general population who are considered to be at high risk of developing lung cancer.

DETAILED DESCRIPTION:
Lung carcinoma is one the most fatal cancer in the world. The enormous fatality rate reflects the limited chance of cure, with a dismal overall 5-year survival rate of approximately 14%. The prognosis of lung cancer depends largely on early detection and immediate treatment prior to metastatic spread. For Stage 1 lung cancer the 5-year survival rate can be as high as 70% . These data suggest that early detection and surgical treatment would have a huge beneficial effect on the lung cancer population. We developed a single arm observational study for the early detection of lung cancer with low dose CT scan in high risk asymptomatic subjects. A mainly non invasive algorithm for management of undetermined nodules was designed including low dose CT at three months for baseline nodules with diameter between 5 and 8 mm, a PET scan for nodules larger that 8 mm (not reduced after antibiotics and one month follow up CT). Lesions increasing in diameter or in density or positive nodules at CT/PET were sent to surgical biopsy (videothoracoscopic approach preferred).

Spirometry was done in all subjects prior to CT scan to evaluate correlation between BPCO and lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50
* Current daily smokers or former smokers (total dose ≥ 20 pack/year, calculated by multiplying the number of packs per day by the total number of years smoked)
* Former smoker should have stopped smoking within the 10 years before the inclusion in the study protocol

Exclusion Criteria:

* Not currently suffering from malignant disease or having had malignant disease within the last 5 years
* Not having known pulmonary pathology
* Not having performed a chest CT scan during the last 2 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 5203 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of malignant pulmonary disease at the first CT examination | once after enrollment
  CT scan
To assess the radiological detection of disease during the 10 year follow-up | once per year for a 10 year follow-up period
  CT scan

SECONDARY OUTCOMES:
To determine the overall resectability of detected malignant tumours | once after detection of malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Bellomi, PhD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Result] Veronesi G, Bellomi M, Mulshine JL, Pelosi G, Scanagatta P, Paganelli G, Maisonneuve P, Preda L, Leo F, Bertolotti R, Solli P, Spaggiari L. Lung cancer screening with low-dose computed tomography: a non-invasive diagnostic protocol for baseline lung nodules. Lung Cancer. 2008 Sep;61(3):340-9. doi: 10.1016/j.lungcan.2008.01.001. Epub 2008 Mar 4. PMID 18308420
- [Result] Pelosi G, Sonzogni A, Veronesi G, De Camilli E, Maisonneuve P, Spaggiari L, Manzotti M, Masullo M, Taliento G, Fumagalli C, Bellomi M, Travis WD, Kadivar M, Viale G. Pathologic and molecular features of screening low-dose computed tomography (LDCT)-detected lung cancer: a baseline and 2-year repeat study. Lung Cancer. 2008 Nov;62(2):202-14. doi: 10.1016/j.lungcan.2008.03.012. Epub 2008 May 2. PMID 18450320
- [Result] Veronesi G, Bellomi M, Veronesi U, Paganelli G, Maisonneuve P, Scanagatta P, Leo F, Pelosi G, Travaini L, Rampinelli C, Trifiro G, Sonzogni A, Spaggiari L. Role of positron emission tomography scanning in the management of lung nodules detected at baseline computed tomography screening. Ann Thorac Surg. 2007 Sep;84(3):959-65; discussion 965-6. doi: 10.1016/j.athoracsur.2007.04.058. PMID 17720408